CLINICAL TRIAL: NCT06087601
Title: The Impact of Genicular Nerves Chemical Neurolysis on the Quality of Life of Patients with Advanced Knee Osteoarthritis. a Randomized, Double-blinded, Clinical Trial
Brief Title: The Impact of Genicular Nerves Chemical Neurolysis on the Quality of Life of Patients with Advanced Knee Osteoarthritis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6/2023
Record Dates: First submitted 2023-07-05; First posted 2023-10-18 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-03

CONDITIONS: Osteo Arthritis Knee; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Sodium Chloride; Ethanol

STUDY DESIGN:
Intervention Model Description: Group 1: sham blocks Group 2: genicular nerve neurolysis
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham blocks (Active Comparator): US-guided Bilateral genicular nerve block with 0,9% NaCl
  Interventions: Drug: 0.9% Sodium chloride
- Genicular nerve neurolysis (Active Comparator): US-guided Bilateral genicular nerve neurolysis with 0,5ml 95% ethanol
  Interventions: Drug: 95% ethanol

INTERVENTIONS:
Drug: 0.9% Sodium chloride — us-guided bilateral genicular nerves sham block with 0,5ml 0,9% normal saline
  Other Names: Sham block
  Arms: Sham blocks
Drug: 95% ethanol — us-guided bilateral genicular nerves neurolysis with 0,5ml 95% ethanol
  Other Names: neurolisis
  Arms: Genicular nerve neurolysis

SUMMARY:
Genicular nerves chemical neurolysis in advanced osteoarthritis of the knee joint.

DETAILED DESCRIPTION:
The study aims to assess the safety and effectiveness of regional pain treatment methods and their impact on the quality of life of patients with advanced osteoarthritis of the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Pain Treatment Clinic of the Transfiguration of Jesus Clinical Hospital of the Medical University of Poznań will be qualified for the study
* patients with gonarthrosis who failed to achieve satisfactory pain control (NRS>3) despite the use of NSAIDs, Paracetamol, and co-analgesics
* Age of patients: from 18 to 110 years of age.
* Caucasian patients can give informed, complete, written consent.

Exclusion Criteria:

* suspected or diagnosed opioid dependence syndrome
* active cancer
* dementia

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
NRS | 7 days after procedure
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS | 30 days after procedure
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS | 3 months after procedure
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS | 6 months after procedure
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
Health Questionnaire (EQ-5D-5L) | 7 days after surgery
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Health Questionnaire (EQ-5D-5L) | 30 days after surgery
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Health Questionnaire (EQ-5D-5L) | 3 months after surgery
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Health Questionnaire (EQ-5D-5L) | 6 months after surgery
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
neurological deficits | 7 days after procedures
  yes/no
neurological deficits | 30 days after procedures
  yes/no
neurological deficits | 3 months after procedures
  yes/no
neurological deficits | 6 months after procedures
  yes/no
total opioid consumption | 7 days after procedure
  milligrams of oral morphine per day
total opioid consumption | 30 days after procedure
  milligrams of oral morphine per day
total opioid consumption | 3 months after procedure
  milligrams of oral morphine per day
total opioid consumption | 6 months after procedure
  milligrams of oral morphine per day

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Wieczorowska-Tobis, Prof.dr hab, Study Director — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No